CLINICAL TRIAL: NCT01769989
Title: Evaluation of the Safety and Efficacy of Electrodermabrasion in Improving the Appearance of Scars That Result From Dermatologic Surgery Compared to Treatment With Dermabrasion
Brief Title: Electrodermabrasion Compared to Dermabrasion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 259842
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Scar
MeSH Terms: conditions — Cicatrix | interventions — Dermabrasion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eletrodermabrasion (Active Comparator): The side treated with electrodermabrasion will be burned with an electric cautery machine to remove the outermost layer of skin as well as the lumps and bumps and a small area of surrounding skin.
  Interventions: Procedure: Electrodermabrasion
- Dermabrasion (Active Comparator): The side treated with dermabrasion will be scraped with a sterile piece of sandpaper until the outermost layer of skin and lumps and bumps have been removed and a small layer of surround skin.
  Interventions: Procedure: Dermabrasion

INTERVENTIONS:
Procedure: Electrodermabrasion
  Arms: Eletrodermabrasion
Procedure: Dermabrasion
  Arms: Dermabrasion

SUMMARY:
The purpose of this study is to determine if electrodermabrasion improves the cosmetic appearance of raise or bumpy scars or scars that are a different color or texture than the surrounding skin resulting from dermatologic surgery and whether it is as good as to the already used method of dermabrasion.

ELIGIBILITY:
Inclusion Criteria:

* Not incarcerated
* No mental impairments that could potentially interfere with the subject's ability to understand the various scar revision modalities and their potential risks and benefits, and thereby ability to provide informed consent
* No bleeding disorders
* A patient at UC Davis Medical Center's Department of Dermatology who has undergone a dermatologic surgery procedure and is not satisfied with the appearance of his/her scar

Exclusion Criteria:

* Incarcerated
* With mental impairment(s) that could potentially interfere with subject's ability to understand the various scare revision modalities and their potential risks and benefits, and thereby ability to provide informed consent
* With a bleeding disorder
* With any other contraindication to the treatment used in the study
* Not a patient at UC Davis Medical Center's Department of Dermatology
* Subjects who are not willing or able to return for follow-up assessments
* Subjects who are not able to give informed consent to enter the study
* Subjects who are not willing to complete the visual analog scale following treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Electrodermabrasion compared to dermabrasion | 3 months
  To determine if electrodermabrasion improves the cosmetic appearance of scars that result from dermatologic surgery better than the current method of dermabrasion.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis, Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical